CLINICAL TRIAL: NCT00000651
Title: A Randomized, Double Blind, Comparative Study of Dideoxycytidine (ddC) Alone or ddC/AZT Combination Versus Zidovudine (ZDV) Alone in Patients With HIV Infection Who Have Received Prior ZDV Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Hoffmann-La Roche (Industry); Glaxo Wellcome (Industry)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 155; 11130 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Zalcitabine; Antiviral Agents; Zidovudine
MeSH Terms: conditions — HIV Infections | interventions — Zidovudine; Zalcitabine

INTERVENTIONS:
Drug: Zidovudine
Drug: Zalcitabine

SUMMARY:
To evaluate the safety of zalcitabine (dideoxycytidine; ddC) alone and in combination with zidovudine (AZT) versus AZT alone when administered to asymptomatic patients with a CD4 count = or < 200 cells/mm3 and symptomatic patients with a CD4 count = or < 300 cells/mm3. To compare the effectiveness of ddC alone and in combination with AZT versus AZT alone.

ddC has been shown to demonstrate an antiviral effect. AZT has been shown to significantly decrease mortality and reduce the frequency of opportunistic infections in patients with AIDS or advanced ARC. After 1 year of AZT therapy, the effectiveness tends to diminish and patients progress with more opportunistic infections and higher mortality rates. Because of the demonstrated antiviral activity, absence of hematologic toxicity, and lack of cross tolerance in laboratory studies of ddC, a study to investigate the long-term effectiveness of ddC in patients with HIV infection who have received AZT therapy is warranted.

DETAILED DESCRIPTION:
ddC has been shown to demonstrate an antiviral effect. AZT has been shown to significantly decrease mortality and reduce the frequency of opportunistic infections in patients with AIDS or advanced ARC. After 1 year of AZT therapy, the effectiveness tends to diminish and patients progress with more opportunistic infections and higher mortality rates. Because of the demonstrated antiviral activity, absence of hematologic toxicity, and lack of cross tolerance in laboratory studies of ddC, a study to investigate the long-term effectiveness of ddC in patients with HIV infection who have received AZT therapy is warranted.

Patients are randomly assigned to 1 of 3 treatment groups. In study arm 1, patients receive AZT plus ddC placebo. In study arm 2, patients receive ddC plus AZT placebo capsules. In study arm 3, patients receive ddC plus AZT. Patients are seen every other week for first 8 weeks and monthly thereafter. Patients are stratified by HIV disease status, length of time receiving AZT, and systemic or local Pneumocystis carinii pneumonia (PCP) prophylaxis. Patients who reach a clinical AIDS-defining endpoint are offered open-label combination therapy.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Required:

* Zidovudine (AZT) = or > 300 mg/day for 6 weeks prior to study entry.

Allowed:

* Chemoprophylaxis for Pneumocystis carinii pneumonia (PCP), candidiasis, and herpes.
* 21 day course of adjuvant systemic corticosteroids for moderate to severe PCP.
* Maintenance treatment with pyrimethamine, sulfadiazine, amphotericin, fluconazole, ketoconazole, acyclovir, ganciclovir, or medications for tuberculosis or Mycobacterium avium for patients who have recovered from toxoplasmosis, cryptococcosis, candidiasis, herpes virus infections, cytomegalovirus infections, tuberculosis or Mycobacterium avium intracellulare.
* 14 day course of metronidazole.
* Erythropoietin and megace if clinically indicated.
* Isoniazid if patient has no peripheral neuropathy at entry and is taking pyridoxine = or > 50 mg/day concomitantly.
* Phenytoin if patient has < grade 2 peripheral neuropathy at entry and has been stable on phenytoin = or > 3 months.

Patients must have:

* Ability and willingness to give informed consent.
* Written informed consent from a parent or guardian if < 18 years old.
* Been tolerating zidovudine (AZT) therapy.
* Diagnosis of HIV infection.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Kaposi's sarcoma or other malignancy requiring therapy.
* Active opportunistic infections.
* Peripheral neuropathy as manifested by complaints of moderate pain, burning, numbness, or tingling in hands/arms or feet/legs; moderate sensory deficit in the upper or lower extremities; or motor weakness in the upper or lower extremities.

Concurrent Medication:

Excluded:

* Other experimental medications.
* Other anti-HIV drugs.
* Biologic response modifiers.
* Cytotoxic chemotherapy.
* Drugs that could cause peripheral neuropathy including phenytoin not specifically allowed, hydralazine, nitrofurantoin, vincristine, cisplatinum, dapsone, disulfiram, and diethyldithiocarbamate.

Concurrent Treatment:

Excluded:

* Radiation therapy.

Patients with the following are excluded:

* Active opportunistic infection. Must have ended acute therapy at least 14 days prior to study entry.
* Peripheral neuropathy = or > grade 2.
* History of intolerance to 500 to 600 mg/day of zidovudine (AZT) as manifested by the same recurrent grade 3 toxicity requiring dose interruptions and dose reductions to < 500 mg/day or any prior grade 4 toxicity.
* Prior development of peripheral neuropathy on ddI = or > grade 2.

Prior Medication:

Excluded:

* Dideoxycytidine (ddC).

Required:

* Zidovudine (AZT) for total of at least 24 weeks; and included within that time period, AZT = or > 300 mg/day for 6 weeks prior to the study entry.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 750
Dates: Study Completion 1993-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M Fischl, Study Chair; A Collier, Study Chair
Locations (40):
- United States (40):
  - USC CRS, Los Angeles, California
  - UCLA CARE Center CRS, Los Angeles, California
  - UCSD Maternal, Child, and Adolescent HIV CRS, San Diego, California
  - Ucsd, Avrc Crs, San Diego, California
  - Ucsf Aids Crs, San Francisco, California
  - Harbor-UCLA Med. Ctr. CRS, Torrance, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Northwestern University CRS, Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Tulane Hemophilia Treatment Ctr., New Orleans, Louisiana
  - Tulane Med. Ctr. - Charity Hosp. of New Orleans, ACTU, New Orleans, Louisiana
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - HMS - Children's Hosp. Boston, Div. of Infectious Diseases, Boston, Massachusetts
  - Bmc Actg Crs, Boston, Massachusetts
  - Beth Israel Deaconess - East Campus A0102 CRS, Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - Brigham and Women's Hosp., Div. of Infectious Disease, Boston, Massachusetts
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - St. Louis ConnectCare, Infectious Diseases Clinic, St Louis, Missouri
  - Washington U CRS, St Louis, Missouri
  - NJ Med. School CRS, Newark, New Jersey
  - SUNY - Buffalo, Erie County Medical Ctr., Buffalo, New York
  - NYU Med. Ctr., Dept. of Medicine, New York, New York
  - Cornell University A2201, New York, New York
  - Memorial Sloan-Kettering Cancer Ctr., New York, New York
  - Beth Israel Med. Ctr. (Mt. Sinai), New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Carolinas HealthCare System, Carolinas Med. Ctr., Charlotte, North Carolina
  - Duke Univ. Med. Ctr. Adult CRS, Durham, North Carolina
  - Regional Center for Infectious Disease, Wendover Medical Center CRS, Greensboro, North Carolina
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Case CRS, Cleveland, Ohio
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio
  - Pitt CRS, Pittsburgh, Pennsylvania
  - University of Washington AIDS CRS, Seattle, Washington

REFERENCES:
- [Background] Blum AS, Dal Pan GJ, Feinberg J, Raines C, Mayjo K, Cornblath DR, McArthur JC. Low-dose zalcitabine-related toxic neuropathy: frequency, natural history, and risk factors. Neurology. 1996 Apr;46(4):999-1003. doi: 10.1212/wnl.46.4.999. PMID 8780079
- [Background] Fichtenbaum CJ, Clifford DB, Powderly WG. Risk factors for dideoxynucleoside-induced toxic neuropathy in patients with the human immunodeficiency virus infection. J Acquir Immune Defic Syndr Hum Retrovirol. 1995 Oct 1;10(2):169-74. doi: 10.1097/00042560-199510020-00009. PMID 7552481
- [Background] Fischl M, Collier A, Stanley K, Ardunio JM, Kazial K, Stein D. The safety and efficacy of zidovudine (ZDV) and zalcitabine (ddC) or ddC alone versus ZDV. ACTG 155 Team of the NIAID. Int Conf AIDS. 1993 Jun 6-11;9(1):68 (abstract no WS-B25-1)
- [Background] Keruly J, Kendig N, Feinberg J, Cotton S, Biggs M, Benjamin Y, Francis H, Wade W, Coplin M, Bartlett J. A model for conducting AIDS clinical trials in a state correctional system. Int Conf AIDS. 1992 Jul 19-24;8(2):B236 (abstract no PoB 3873)
- [Background] Johnson VA. Combination therapy: more effective control of HIV type 1? AIDS Res Hum Retroviruses. 1994 Aug;10(8):907-12. doi: 10.1089/aid.1994.10.907. PMID 7811541
- [Background] Fischl MA, Stanley K, Collier AC, Arduino JM, Stein DS, Feinberg JE, Allan JD, Goldsmith JC, Powderly WG. Combination and monotherapy with zidovudine and zalcitabine in patients with advanced HIV disease. The NIAID AIDS Clinical Trials Group. Ann Intern Med. 1995 Jan 1;122(1):24-32. doi: 10.7326/0003-4819-122-1-199501010-00004. PMID 7985892
- [Background] Spino C, Kahn JO, Dolin R, Phair JP. Predictors of survival in HIV-infected persons with 50 or fewer CD4 cells/mm3. J Acquir Immune Defic Syndr Hum Retrovirol. 1997 Aug 15;15(5):346-55. doi: 10.1097/00042560-199708150-00004. PMID 9342254
- [Background] Zackin RA, Clark RA, Currier JS, Mildvan D. Predictive markers of HIV-related weight loss and determination of differences between populations with weight loss stratified by opportunistic processes. J Acquir Immune Defic Syndr. 1999 Oct 1;22(2):189-93. doi: 10.1097/00126334-199910010-00012. PMID 10843534